CLINICAL TRIAL: NCT00053963
Title: A PHASE I STUDY OF DEPSIPEPTIDE (NSC#630176, IND# 51810) IN PEDIATRIC PATIENTS WITH REFRACTORY SOLID TUMORS AND LEUKEMIAS
Brief Title: FR901228 in Treating Children With Refractory or Recurrent Solid Tumors or Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01803; ADVL0212; U01CA097452 (NIH); CDR0000269671 (Registry Identifier: PDQ (Physician Data Query)); NCT00069771 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Blastic Phase Chronic Myelogenous Leukemia; Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Chronic Myelogenous Leukemia; Childhood Craniopharyngioma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Spinal Cord Neoplasm; Childhood Supratentorial Ependymoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Blast Crisis; Choroid Plexus Neoplasms; Astrocytoma; Spinal Cord Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — romidepsin

ARMS (1):
- Arm I (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax

SUMMARY:
This phase I trial is studying the side effects and best dose of FR901228 in treating children with refractory or recurrent solid tumors or leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of FR901228 (depsipeptide) in pediatric patients with refractory or recurrent solid tumors.

II. Determine the dose-limiting toxic effects of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Assess tolerability of this drug at the solid tumor MTD in patients with refractory or recurrent leukemia.

V. Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients with solid tumors receive escalating doses of FR901228 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Cohorts of 3 patients (6 patients total) with leukemia receive FR901228 as above at the MTD.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy

  * Extracranial solid tumors or brain tumors*
  * Diagnosis of leukemia allowed after maximum tolerated dose is determined, including any of the following:

    * Acute lymphoblastic leukemia
    * Acute myelogenous leukemia
    * Chronic myelogenous leukemia in blast crisis
* Disease must be refractory to conventional therapy or no effective conventional therapy exists
* CNS tumors resulting in neurological deficits must be stable for 2 weeks before study entry
* Performance status - Karnofsky 60-100% (over 10 years old)
* Performance status - Lansky 60-100% (10 years old and under)
* At least 8 weeks
* Absolute neutrophil count at least 1,000/mm^3 (for solid tumor patients without bone marrow involvement)
* Platelet count at least 100,000/mm^3 (for solid tumor patients without bone marrow involvement; platelet transfusion independent) OR 20,000/mm^3 (for leukemia patients; platelet transfusion allowed)
* Hemoglobin at least 8.0 g/dL (RBC transfusions allowed)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 5 times ULN
* Albumin at least 2 g/dL
* Glomerular filtration rate at least 70 mL/min
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (for patients 5 years of age and under)
  * No greater than 1.0 mg/dL (for patients 6 to 10 years of age)
  * No greater than 1.2 mg/dL (for patients 11 to 15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)
* Calcium normal (with or without supplementation)
* Shortening fraction at least 27% by echocardiogram OR ejection fraction at least 50% by MUGA
* No symptomatic congestive heart failure
* No uncontrolled cardiac arrhythmia
* QTc less than 450 msec
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry greater than 94%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study treatment
* Magnesium and potassium normal (with or without supplementation)
* No uncontrolled seizure disorder
* No uncontrolled infection
* No graft-vs-host disease
* No seizure disorder unless well controlled and not on enzyme-inducing anticonvulsants
* At least 1 week since prior growth factors
* At least 3 weeks since prior biologic therapy or immunotherapy and recovered
* At least 6 months since prior allogeneic stem cell transplantation
* No concurrent routine prophylactic growth factors
* At least 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No prior FR901228 (depsipeptide)
* No other concurrent anticancer chemotherapy
* Concurrent dexamethasone for CNS tumors allowed if on stable dose or decreasing dose for at least 1 week before study entry
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior craniospinal radiotherapy or radiotherapy to at least 50% of pelvis
* At least 6 weeks since other prior substantial bone marrow radiation
* More than a 5 half-life washout period since prior and no concurrent medications associated with prolongation of QTc interval
* No concurrent enzyme-inducing anticonvulsants
* No concurrent hydrochlorothiazide
* No other concurrent investigational drugs

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2002-09; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
MTD, defined as that dose at which fewer than one-third of patients experience DLT, graded according to the NCI CTC version 2.0 | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States